CLINICAL TRIAL: NCT03770884
Title: Rheumatism and Dietetic: RHUMADIET Study (Food Practices and Beliefs)
Acronym: RHUMADIET
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18027J; 2018-A01340-55 (Other: ANSM); HAO18041 (Other Grant/Funding Number: Association)
Record Dates: First submitted 2018-07-09; First posted 2018-12-10 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis; Axial Spondyloarthritis; Hand Osteoarthritis
Keywords: rheumatoid arthritis; Axial spondyloarthritis; hand osteoarthritis; diet; beliefs
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis: EULAR-ACR criteria Whatever the treatment and the disease activity
- Axial spondyloarthritis: ASAS criteria for axial disease Whatever the treatment and the disease activity
- digital osteoarthritis: According to ACR criteria Whatever the treatment and the disease activity

SUMMARY:
Cross sectional study assessing food practices and beliefs in RA, AS and DA (digital arthritis)

DETAILED DESCRIPTION:
To investigate in patients having rheumatoid arthritis (RA), or axial spondyloarthritis (AS) or digital osteoarthritis (DA) practices and beliefs about influence of food and diet on their rheumatic disease.

200 patients of each disease will be included in this cross-sectional non interventional study Factors associated with specific practices or specific beliefs will be determined.

Only questionnaires are used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Rheumatoid arthritis (RA) according to ACR/EULAR criteria or axial spondyloarthritis (AS) according to ASAS 2009 criteria or digital osteoarthritis (DA) according to ACR criteria.

Exclusion Criteria:

* Severe upper functional or psychiatric disorders
* Patients under guardianship or trusteeship
* Patients unable to answer the questionnaire in French

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA (EULAR/ACR criteria) AS (ASAS criteria ) DA (ACR criteria)
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who follow or have followed at least one diet for their rheumatic disease among gluten-free, cow's milk, lactose-free, vegetarian, vegan, Seignalet, Mediterranean, fasting period | 10 minutes
  Binary criterion: Diet follower Yes/No

SECONDARY OUTCOMES:
comparison between each rheumatism rheumatoid arthritis, Axial spondyloarthritis digital osteoarthritis of the prevalence of patients having followed or following one or more diets | 10 minutes
  Proportion of diet follower patients in RA versus AS versus DA. Specific food and diet questionnaires will be used in this study.
For each type of food, prevalence of patients with RA considering that the food influences the rheumatic pain in each rheumatic disease | 10 minutes
  for each type of food (meat, vegetables, fruits, grains, nuts, fish, alcohol, soda), prevalence of patients with RA considering that food influence their disease symptoms
For each type of food, prevalence of patients with AS considering that the food influences the rheumatic pain in each rheumatic disease | 10 minutes
  for each type of food (meat, vegetables, fruits, grains, nuts, fish, alcohol, soda), prevalence of patients with AS considering that food influence their disease symptoms
For each type of food, prevalence of patients with DA considering that the food influences the rheumatic pain in each rheumatic disease | 10 minutes
  for each type of food (meat, vegetables, fruits, grains, nuts, fish, alcohol, soda), prevalence of patients with DA considering that food influence their disease symptoms
Research of socio-demographic or rheumatic factors associated with dieting in RA. | 10 minutes
  In RA population:Unajusted and adjusted risk of diet (odds ratio) assiociated with the following factors reported from patient file or patient questionnaires.
  * Sociodemorgraphic parameters:Age, gender, education level.
  * Physiologic parameters: Autoantibody status, BMI
  * Clinical parameters: treatments, disease activity using DAS 28 scale.
Research of socio-demographic or rheumatic factors associated with dieting in AS. | 10 minutes
  In AS population: Unajusted and adjusted risk of diet (odds ratio) assiociated with the following factors reported from patient file or patient questionnaires.
  * Sociodemorgraphic parameters:Age, gender, education level.
  * Physiologic parameters: BMI
  * Clinical parameters: treatments, disease activity using BASDAI Scale
Research of socio-demographic or rheumatic factors associated with dieting in DA. | 10 minutes
  In DA population: Unajusted and adjusted risk of diet (odds ratio) assiociated with the following factors reported from patient file or patient questionnaires.
  * Sociodemorgraphic parameters: Age, gender, education level.
  * Physiologic parameters: BMI
  * Clinical parameters: treatments, disease activity using 0-100mm visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie SELLAM, Prof,MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rhumatologie - Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No